CLINICAL TRIAL: NCT01497262
Title: A 4-month, Open-label, Multi-center Study to Explore the Safety and Tolerability of Fingolimod 0.5 mg in Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: Safety and Tolerability of Fingolimod in Patients With Relapsing-remitting Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720D2325
Record Dates: First submitted 2011-12-05; First posted 2011-12-22 (Estimated); Results first posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fingolimod Hydrochloride

ARMS (1):
- Fingolimod (Experimental): Open-label fingolimod 0.5 mg, taken orally once daily for 4 months
  Interventions: Drug: Fingolimod

INTERVENTIONS:
Drug: Fingolimod — Fingolimod will be supplied as 0.5mg capsules in bottles of 35.

SUMMARY:
This 4 month, open-label study will evaluate the safety and tolerability of fingolimod 0.5 mg in patients with relapsing-remitting multiple sclerosis (RRMS) and generate additional data in Multiple Sclerosis (MS) patient population that closely resembles the clinical population seen in routine medical care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsing remitting Multiple Sclerosis
* Patients with Expanded Disability Status Scale (EDSS) score of 0-6.5.

Exclusion Criteria:

* Patients with MS other than relapsing remitting MS
* Patients with a history of chronic disease of the immune system other than MS, which requires systemic immunosuppressive treatment, or a known immunodeficiency syndrome.
* Patients who have been treated with:

  * systemic corticosteroids or immunoglobulins within 1 month prior to baseline;
  * immunosuppressive medications within 3 months prior to baseline;
  * monoclonal antibodies within 3 months prior to baseline;
  * cladribine, mitoxantrone or alemtuzumab at any time.
* Uncontrolled diabetes mellitus at screening
* Diagnosis of macular edema during Screening Phase
* Patients with active systemic bacterial, viral or fungal infections, or known to have AIDS, Hepatitis B, Hepatitis C infection or to have positive HIV antibody, Hepatitis B surface antigen or Hepatitis C antibody tests.
* Patients who have received total lymphoid irradiation or bone marrow transplantation.
* Patients with certain cardiovascular conditions and/or findings in the screening ECG
* Patients with certain liver conditions
* Pregnant confirmed by a positive pregnancy test t or nursing (lactating) women
* Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2012-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (24):
- Argentina (5):
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Villa Nueva, Mendoza Province
  - Novartis Investigative Site, Salta, Salta Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Córdoba
- Brazil (2):
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
- Colombia (4):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Bogotá, Cundinamarca
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Cali
- Jordan (2):
  - Novartis Investigative Site, Amman, Amman Governorate
  - Novartis Investigative Site, Irbid
- Malaysia (3):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, George Town, Pulau Pinang
  - Novartis Investigative Site, Kuala Lumpur
- Mexico (4):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, San Nicolás de los Garza, Nuevo León
  - Novartis Investigative Site, San Luis Potosí City, San Luis Potosí
- Novartis Investigative Site, Panama City, Provincia de Panamá, Panama
- Peru (3):
  - Novartis Investigative Site, Jesus Maria, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, La Perla, Provincia Constitucional del Callao

REFERENCES:
- [Derived] Ordonez-Boschetti L, Rey R, Cruz A, Sinha A, Reynolds T, Frider N, Alvarenga R. Safety and Tolerability of Fingolimod in Latin American Patients with Relapsing-Remitting Multiple Sclerosis: The Open-Label FIRST LATAM Study. Adv Ther. 2015 Jul;32(7):626-35. doi: 10.1007/s12325-015-0224-2. Epub 2015 Jul 14. PMID 26170105

RESULTS

PARTICIPANT FLOW:
Groups:
- Fingolimod 0.5 mg: Open-label fingolimod 0.5 mg, taken orally once daily for 4 months
Period: Overall Study
Arm/Group | Fingolimod 0.5 mg
Started | 162
Completed | 151
Not Completed | 11
Not completed — Abnormal Lab Values | 4
Not completed — Abnormal Test Procedure Result | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: The Enrolled Set (ENR) included all patients who signed the informed consent and enrolled in study
Arm/Group | Fingolimod 0.5 mg
Number analyzed (Participants) | 162
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.3 (9.67)
Age, Customized [Number; unit: Participants]
  <18 years | 0
  18-30 years | 47
  31-40 years | 60
  41-55 years | 47
  56-65 years | 8
  >65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114
  Male | 48

OUTCOME MEASURES:

1. Secondary Outcome: Number (%) of Patients With AE of Special Interest Including Bradyarrhythmia, BP Increase, Liver Transaminase Elevations, Infections , Macula Oedema.
Description: The incidence of events in special areas of safety interest (including bradyarrhythmias, BP increase, liver function, infections and macular oedema) were assessed by the nature and frequency of AE reporting. These areas of special interest have been identified and potential risks of fingolimod based on knowledge from clinical trials and post-marketing reporting.
Time Frame: 4 months
Population: Safety set includes all patients who received at least one dose of study drug
Measure: Number; unit: Percent of Participants
Arm/Group | Fingolimod 0.5 mg
Number analyzed (Participants) | 162
Percent of Participants
  Bradyarrhythmias | 8.6
  Blood pressure increase | 0.6
  Hypertension | 2.5
  Liver Transaminase evaluations | 3.7
  Infections | 28.4
  Macula Oedema | 0

2. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Any Adverse Event was defined as occurrence of any symptom regardless of intensity grade, Serious Adverse Event (SAEs) assessed as medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in persistent or significant disability/incapacity
Time Frame: 28 weeks
Population: Safety set includes all patients who received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Fingolimod 0.5 mg
Number analyzed (Participants) | 162
Participants
  Adverse Events (AE) | 100
  Serious Adverse Event (SAE) | 12
  Deaths | 0

ADVERSE EVENTS:
Time Frame: Weeks 2,8, 16 and end of study visit
Description: Safety set includes all patients who took at least one dose of study drug
Arm/Group | Fingolimod 0.5 mg
Serious Adverse Events (participants affected / at risk) | 12/162
Other Adverse Events (participants affected / at risk) | 63/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod 0.5 mg (N=162)
Leukopenia (Blood and lymphatic system disorders) | 1
Gastroenteritis (Infections and infestations) | 2
Gastroenteritis viral (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fibrin D dimer increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Multiple sclerosis relapse (Nervous system disorders) | 3
Optic neuritis (Nervous system disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod 0.5 mg (N=162)
Lymphopenia (Blood and lymphatic system disorders) | 17
Bradycardia (Cardiac disorders) | 6
Vision blurred (Eye disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 10
Influenza (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 22
Anxiety (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.